CLINICAL TRIAL: NCT01958502
Title: Evaluation the Treatment of Nonunion of Long Bone Fracture of Lower Extremities (Femur and Tibia) Using Mononuclear Stem Cells From the Iliac Wing Within a 3-D Tissue Engineered Scaffold
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Emdadi Kamyab Hospital (Other)
Collaborators: National Taiwan University of Science and Technology (Other)
Responsible Party: Principal Investigator, mohammad taghi peivandi, MD, Emdadi Kamyab Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 910359
Record Dates: First submitted 2013-08-21; First posted 2013-10-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Nonunion of Fracture
Keywords: nonunion; mesenchymal stem cell; scaffold; BMP2; long bone
MeSH Terms: conditions — Fractures, Ununited

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mesenchymal stem cell (Experimental): stem cells drived from iliac bone marrow with centrifuge and ficoll method then implant in collagenic 3-D scaffold with BMP-2 and put in non union site by surgical approach under general or spinal anesthesia as deemed appropriate by the anesthetist.
  Interventions: Genetic: surgical treatment of non union with mesenchymal stem cells with BMP2 within a 3-D tissue engineered scaffold

INTERVENTIONS:
Genetic: surgical treatment of non union with mesenchymal stem cells with BMP2 within a 3-D tissue engineered scaffold

SUMMARY:
Because the rate of non union of long bone in lower extremities specially in tibia in this two last decade due to malnutrition and smoking and other risk factors was increased, so many patient in our country suffer from non union. On the other hand it seems that the use of the mesenchymal stem cells can irritate the union rate. Also for better result we used the mesenchymal stem cells with BMP2 in collagenic scaffold. The collagen has a osteoconductive effect and BMP2 and stem cells has a osteoinductive effect therefore this combination is useful in filling the gap in non union site and irritate the union rate.

Mesenchymal stem cell derived from iliac bone marrow after centrifuge with ficoll procedure. Then the investigators will follow the patient with monthly radiography and evaluate the callus volume and clinical union and any side effect of this treatment. Clinical union consider to relief pain in non union site and be stable in examination.

ELIGIBILITY:
Inclusion Criteria:

* Every patient with non union in the site of long bone fracture
* Age more than 18 and under 60 years old
* Fracture having no radiological callus after 6 months and absence of any hypertrophic bone reaction.
* No infection in site of surgery
* Be able and willing to participate in the study
* Written informed consent

Exclusion Criteria:

* Evidence of malignancy
* Pregnancy or breastfeeding
* Patient positive by serology or PCR for HIV, hepatitis B or C infection the patient with Accompanied fracture such as hip fracture that could not weight bearing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
clinical and radiological union at 1 month to 6 months | 6 months
  patients receiving Mesenchymal Stem Cells within a 3-D tissue engineered scaffold that develop a partial or complete callus at 1, 2, 3, 4 ,5 and 6 months evaluate with standard X-rays

SECONDARY OUTCOMES:
Safety of Mesenchymal Stem Cells injection in nonunion fractures. Follow-up for revealing any significant immediate or late adverse effects(infection,malignancy,local or systemic allergic reaction) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: mohammad taghi peivandi, MD, Principal Investigator — Emdadi Kamyab Hospital; amin razi, MD, Study Director — Emdadi Kamyab Hospital
Locations (1):
- Emdai Kamyab Hospital, Mashhad, Khorasan, Iran